CLINICAL TRIAL: NCT04787939
Title: Early Feeding After Free Flap Reconstruction of Oral Cavity Defects: A Single Arm Non-inferiority Trial
Brief Title: Early Feeding After Oral Cavity Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Mohemmed Khan, Assistant Professor, Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HSM 20-01801
Record Dates: First submitted 2021-03-04; First posted 2021-03-09 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Head and Neck Cancer; Free Tissue Transfer
Keywords: Oral Cavity Cancer; Oral Cavity Reconstruction; Early Postoperative Feeding; Orocutaneous Fistula; Salivary Leak
MeSH Terms: conditions — Head and Neck Neoplasms; Mouth Neoplasms

STUDY DESIGN:
Intervention Model Description: The study is a single arm non-inferiority study evaluating wound healing outcomes (orocutaneous fistula, salivary leak, wound dehiscence) in subjects undergoing free tissue transfer for oral cavity reconstruction who are permitted to drink liquids by mouth on postoperative day 1. Outcomes are tracked and assessed over a 30 day period postoperatively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early Feeding Arm (Experimental): Early Feeding Group
  Interventions: Behavioral: Early Feeding

INTERVENTIONS:
Behavioral: Early Feeding — Subjects will be permitted to drink liquids by mouth on the first day after surgery. Outcomes related to their care, wound healing, and quality of life will be followed for 30 days after surgery.

SUMMARY:
This is a prospective single-arm non-inferiority trial evaluating surgical outcomes in subjects who are fed in the first days after oral cavity reconstructive surgery. The purpose of the study is to specifically compare the rates of orocutaneous fistula in subjects who are allowed to eat immediately after surgery to those rates published in the literature (individuals for whom oral feeding is delayed for several days after surgery). Eighty nine subjects who will undergo oral cavity reconstructive surgery will be enrolled between Mount Sinai Hospital and Mount Sinai West. Study participation will last for 30 days after surgery during which time patients will be examined for any signs or symptoms of surgical site infection or wound breakdown, have several clinical evaluations of swallow function, and be asked to report on several patient reported outcome measures.

DETAILED DESCRIPTION:
In this single-arm non-inferiority study, the study team will aim to evaluate the safety of early feeding in patients with oral cavity reconstruction who are allowed to eat by mouth on post-operative day 1. Traditionally, surgeons have opted to delay the time to oral feeding in oral cavity reconstruction because of concern that an early oral diet may stress intraoral suture lines and lead to the development of salivary leaks. However, evidence from small studies evaluating oral feeding timing in patients who underwent total laryngectomy suggests that there is no increased risk associated with early oral feeding. As such, the study team will aim to determine whether early feeding on postoperative day 1 is non-inferior with respect to the development of orocutaneous fistula to the standard care as described in the literature. There are roughly 50-60 oral cavity reconstructive surgeries performed at Mount Sinai each year - as such it is not feasible to recruit two study arms for direct comparison.

In addition to salivary leak rates, the study team will report outcomes related to the cohort's wound healing, length of time in the hospital, length of time requiring an enteral tube feeds, swallow evaluation information, and the results of patient reported outcomes measures.

ELIGIBILITY:
Inclusion Criteria

* Patients receiving free tissue transfer regardless of the indication for oral cavity reconstruction will be included.
* Age ≥ 18 years.
* English, Spanish, and Chinese (Mandarin) speaking patients
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria

* Patients having undergone prior major oral cavity surgery or radiation to the oral cavity (also known as surgical salvage patients).
* Patients with a known history of dysphagia or with current enteral feeding needs
* Patients with a history of traumatic brain injury, stroke, or dementia
* Patients unable to understand the research protocol and/or provide informed consent. The consent will be translated into English, Spanish, and Chinese (Mandarin). Given patient demographics at Mount Sinai Hospital, this will include the overwhelming majority of patients.
* Patients under the age of 18
* Patients whose participation in this trial would require exclusion from participation in another clinical research trial related to the patient's malignant diagnosis.
* Vulnerable populations (adults unable to consent, individuals who are not yet adults, wards of the state, pregnant women, prisoners, pregnant women)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Orocutaneous Fistula | 30 days
  Orocutaneous Salivary Fistula Formation - An orocutaneous fistula or salivary leak is a wound complication that results when saliva or other liquids leak from the mouth through the skin of the face or neck. The subject's oral cavity and neck will be monitored in the standard fashion for development of orocutaneous fistula. The oral cavity will be monitored daily for signs of wound breakdown. The neck will be examined for redness, tenderness to palpation, or increased swelling. Additionally, systemic signs of fistula formation will be monitored such as leukocytosis and fever.

SECONDARY OUTCOMES:
Incidence of Surgical Site Infection | 30 days
  Surgical site infection is defined clinically as fever, erythema, swelling or purulent drainage from the surgical site requiring topical or systemic treatment.
Incidence of Wound Dehiscence | 30 days
  Wound dehiscence is defined as the breakdown at the surgical site with or without intervention.
Rate of PO tolerance | 30 days
  The proportion of patients that are cleared for a diet by the speech language pathology team.
Incidence of Aspiration pneumonia | 30 days
  Aspiration pneumonia is defined clinically based on vital signs, respiratory secretions, and chest x-ray findings indicating pneumonia requiring antibiotic treatment.
Length of hospital stay | 30 days
  Length of hospital stay is defined as the days from admission to discharge.
Jaw range of motion | 30 days
  Bedside swallow evaluation outcomes include jaw Jaw Range of Motion opening which will be measured in millimeters using the Therabite measuring tool and fingers, ranges from 0, indicating <1, to 5, indicating 3 or greater.
Tongue range of motion | 30 days
  Bedside swallow evaluation outcomes include tongue range of motion. Tongue Range of Motion Scale will be measured in millimeters, with a range of 100-0, 100 indicating full tongue range of motion and 0 indication no tongue movement.
MD Anderson Dysphagia Index (MDADI) | 30 Days
  MD Anderson Dysphagia Index (MDADI) is a survey designed to assess a subject's perception of his or her swallowing ability. Patient responds to questionnaire that best reflects their current experience, ranges from Strongly Agree to Strongly Disagree. The scores range from a minimum of 0 to a max of 100, with higher scores indicating higher functioning.
Performance Status Scale for Head and Neck Cancer (PSS-HN) | 30 Days
  Performance Status Scale for Head and Neck Cancer (PSS-HN) is a survey aimed at evaluating performance and function with regard to eating, speaking, and eating in public. Subscales provide a range of 100 - No restrictions and full understandability to 0 - Full restrictions and no understandability. Subscales are scored individually with higher scores indicating better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Mohemmed Khan, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Health System, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No